CLINICAL TRIAL: NCT03035422
Title: Sequential Chemotherapy Prior to Reduced Intensity Conditioning: Interventional Study in Haploidentical Hematopoietic Stem Cells Transplantation for Patients With Refractory Acute Myeloid Leukemia
Brief Title: Sequential Conditioning in Haploidentical Transplantation for Refractory Acute Myeloid Leukemia
Acronym: SET-HAPLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A00862-49
Record Dates: First submitted 2016-11-24; First posted 2017-01-30 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Refractory Acute Myeloid Leukemia
Keywords: Allogenic cell stem transplant, Sequential chemotherapy Haploidentical transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with primary refractory acute myeloid leukemia (Other): Patients with primary refractory acute myeloid leukemia
  Interventions: Drug: Sequential Packaging (SET); Drug: Transfusion graft; Drug: Prevention of GVHD; Drug: Care supports; Drug: Lymphocyte injection of prophylactic donor (PDLI)

INTERVENTIONS:
Drug: Sequential Packaging (SET) — Sequential chemotherapy:
  * Thiotepa 5 mg / kg / day for 1 day (D-13)
  * Cyclophosphamide 400 mg / m² / day for 4 days (J-12 to J-9)
  * Etoposide 100 mg / m² / day for 4 days (J-12 to J-9) Repos days J-8 and J-6 Reduced-intensity conditioning (RIC)
  * Fludarabine 30 mg / m² / day for 5 days (J-5 to D-1)
  * Busulfan IV 3.2 mg / kg / day for 2 days (J-5 and J-4)
  * Anti-lymphocyte serum (Thymoglobuline) 2.5 mg / kg / day for 2 days (J-3 and J-2)
Drug: Transfusion graft — Graft of peripheral stem cells is preferred at D0
Drug: Prevention of GVHD — * Cyclophosphamide 50mg / kg / day on days D + 3 and D + 5
  * Cyclosporine A (CSA; 3 mg / kg / day IV from D + 6)
  * Mycophenolate mofetil (MMF; 30 mg / kg / day, maximum x2 1g / day from day J + 6)
Drug: Care supports — According to the protocols of each center
Drug: Lymphocyte injection of prophylactic donor (PDLI) — According to the protocols of each center. In the absence of clinical indication against-disease (GVHD), phasing MMF between days D + 35 and D + 56, then phasing APF between D + 62 and D + 90
  - PDLI: 3 injections from the D + 120 patients who discontinued immunosuppressive therapy for ≥ 1 month and having no active GVHD or history of acute GVHD grade> II

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the only treatment option with a significant chance of healing in acute myeloid leukemia (AML) or refractory multiple relapses after chemotherapy. However, all patients with an indication of allo-HSC can not benefit because of two limitations: the toxicity of the treatment and graft shortage available.

DETAILED DESCRIPTION:
The goal is to evaluate the efficacy and safety of the combination of an SET followed by haploidentical transplant with post-transplant immune modulation by prophylactic DLI in patients with refractory acute myeloid leukemia or relapsed. The main objective is to assess overall survival at 2 years in these patients.

Secondary objectives:

1. To evaluate the efficacy of this therapeutic strategy in terms of remission of disease, incidence of relapse and relapse-free survival
2. To evaluate the non-relapse mortality
3. To evaluate the incidence of acute and chronic graft against host disease (GVHD)
4. To assess the feasibility of prophylactic injections of donor lymphocytes (pDLI)
5. To analyze the post-transplant immune reconstitution

Secondary endpoints:

1. partial or complete remission rate by standard criteria at 90 days and then 6, 12 and 24 months after transplantation.

   Relapse incidence and death related to the disease 90 days 6, 12 and 24 months after transplantation Leukemia-free survival at 1 year and 2 years after transplantation
2. Cumulative incidence of death not related to relapse at 90 days, 1 year and 2 years after transplantation
3. Cumulative incidence of acute and chronic graft against host disease (GVHD)
4. Number of patients for whom pDLI was possible and number of pDLI / patient; incidence, severity and treatment of possible secondary GVHD in these patients
5. Study of immune reconstitution post-transplant in the peripheral blood 30, 90 and 180 days after transplantation (CD4 lymphocyte levels, CD8, T regulators, Natural Killer cells and B cells)

Methodology, experimental design:

Multicenter study in routine care, prospective

All patients will receive, as part of the marketing authorization of the products used, the following regimen:

1- sequential Packaging (SET):

1. sequential chemotherapy:

   * Thiotepa 5 mg / kg / day for 1 day (D-13)
   * Cyclophosphamide 400 mg / m² / day for 4 days (J-12 to J-9)
   * Etoposide 100 mg / m² / day for 4 days (J-12 to J-9)
2. Rest days J-8 and J-6
3. Reduced-intensity conditioning (RIC)

   * Fludarabine 30 mg / m² / day for 5 days (J-5 to D-1)
   * Busulfan IV 3.2 mg / kg / day for 2 days (J-5 and J-4)
   * Anti-lymphocyte serum (Thymoglobuline) 2.5 mg / kg / day for 2 days (J-3 and J-2)

     2 Graft transfusion: the day D0. A graft of peripheral stem cells is preferred.

     3- Prevention of GVHD:
   * Cyclophosphamide 50mg / kg / day on days D + 3 and D + 5
   * Cyclosporine A (CSA; 3 mg / kg / day IV from D + 6)
   * Mycophenolate mofetil (MMF; 30 mg / kg / day, maximum x2 1g / day from day J + 6)

     4- Care supports: according to the protocols of each center

     5- lymphocyte injection of prophylactic donor (pDLI): according to the protocols of each center. The following scheme is proposed:
   * In the absence of clinical contraindication(GVHD), tapering MMF between days D + 35 and D + 56, then tapering CSA between D + 62 and D + 90
   * pDLI: 3 injections from the D + 120 in patients who discontinued immunosuppressive therapy for ≥ 1 month and having no active GVHD or history of acute GVHD grade> II.

     6. Feedback: at baseline and 1, 3, 6, 12 and 24 months after transplant (engraftment, disease response, immune reconstitution, chimerism, GVHD, infection, quality of life).

The treatments evaluated in this strategy are all used in the usual care of patients and follow-up will not be changed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of acute myeloid leukemia after primary induction treatment failure (persistent leukemia after 2 cycles of induction chemotherapy)
* Patient age ≥ 18 to <60 years
* Cardiac ejection fraction of the left ventricle ≥ 45%
* Lung function - free diffusion capacity for carbon monoxide ≥ 50% of predicted value
* Creatinine clearance ≥ 50 ml / min depending on the CKD-EPI formula
* Availability of an HLA haploidentical donor in the family
* Collection of non-opposition

Exclusion Criteria:

* Uncontrolled invasion of CNS
* Availability of an HLA identical family donor who agreed to donate hematopoietic stem cells OR non-related donor HLA-compatible 10/10 on HLA-A alleles, B, C, and DRB1 DQB1 available and ready to give in 4 weeks to make a decision allograft
* Presence in the patient HLA-specific antibodies directed against an antigen HLA haploidentical donor family
* Karnofsky score <70%
* Patient HIV positive
* Hepatitis B or C or chronic active
* Uncontrolled infection at the time of start packing
* Contraindication to the use of treatments provided by the Protocol
* Previous history of allo-HSC
* No beneficiary of a social security scheme.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years after transplantation
  The aim is to describe the efficacy of the combination of a SET followed by haploidentical transplant with post-transplant immune modulation by pDLI in patients with AML.
  The main objective is to assess overall survival at 2 years in these patients.

SECONDARY OUTCOMES:
Partial or complete remission rate by standard criteria Relapse incidence and death related to the disease | 90 days and then 6, 12 and 24 months after transplantation
  To evaluate the efficacy of this therapeutic strategy in terms of remission of disease, incidence of relapse
Cumulative incidence of death not related to relapse | 90 days and then 12 and 24 months after transplantation
  Assess not related to relapse mortality
Cumulative incidence of acute and chronic graft against host disease (GVHD) | 100 days and then 12 and 24 months after transplantation
  To evaluate the incidence of acute and chronic graft against host disease (GVHD)
Number of patients for whom pDLI was possible. | 2 years after transplantation
  Assess the feasibility of prophylactic injections of donor lymphocytes (pDLI)
Study of immune reconstitution post-transplant in the peripheral blood will be used:CD4 lymphocyte levels, CD8, T regulators, Natural Killer cells and B cells | 90 days and then 6, 12 and 24 months after transplantation
  Study the post-transplant immune reconstitution
Leukemia free survival | 90 days and then 6, 12 and 24 months after transplantation
  Relapse-free survival
Number of pDLI / patient; incidence, severity and treatment of possible secondary GVHD in these patients | 90 days and then 6, 12 and 24 months after transplantation
  Assess the feasibility of prophylactic injections of donor lymphocytes (pDLI)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie Clinique Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No